CLINICAL TRIAL: NCT04740463
Title: Assessement of Capacity to Consent in Depressed Patients
Brief Title: Assessement of Capacity to Consent
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0033
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-02

CONDITIONS: Major Depressive Episode
Keywords: Capacity to consent; Euthanasia
MeSH Terms: conditions — Suicide, Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Any patient can request euthanasia in many of our neighbouring European countries as long as informed consent is given. Psychiatric evaluation is not always mandatory.

Faced with the increasing emergence of euthanasia requests in different countries from patients under psychiatric care in France for severe depressive episodes, question arises of a possible alteration in the capacity to give consent in the context of a severe depressive episode.

This is a Social and Human Sciences study which does not aim to modify the usual management of patients.

ELIGIBILITY:
Inclusion criteria:

* Age between 18 and 75
* Ability to understand and participate in the interview
* French-speaking
* Presence of a current characterized depressive episode according to DSM-5 diagnostic criteria

Exclusion criteria:

- Refusal to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Depressed patients (consultation or hospitalization)
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Capacity to consent (MacCAT-T) | 1 day
  aassessment of the capacity to consent based on the MacArthur Competence Assessment Tool-Treatment (MacCAT-T). The questionnaire assesses four competences in consent : understanding (score ranges from 0 to 6), appreciation (score ranges from 0 to 4), reasoning (score ranges from 0 to 8) and expressing a choice (score ranges from 0 to 2).
  A low score on each of these dimensions calls into question the patient's ability to consent.

SECONDARY OUTCOMES:
Insight (BCIS) | 1 day
  insight assessement based on the Beck Cognitive Insight Scale (BCIS). The questionnaire contains two sub-scales : self- reflection (9 items) and self-certainty (6 items). Each items ranges from 0 (do not agree at all) to 3 (agree completely)

OTHER OUTCOMES:
Depression (BDI) | 1 day
  depression assesement based on the Beck Depression Inventory (BDI) score. Total score ranges from 0 to 63. Higher scores indicate more severe depression symptoms.
Depression (MADRS) | 1 day
  depression assessement based on the Montgomery Asberg Depression Rating Scale (MADRS) score. Total score ranges from 0 to 60. Higher scores indicate more severe depression symptoms.
Suicidality (MADRS) | 1 day
  suicidality assessement based on the 10th MADRS item. The item ranges from 0 (enjoys life or takes it as it come) to 6 (explicit plans for suicide when there is an opportunity. Active preparations for suicide).

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Olie, MD PhD, Study Director — University Hospital, Montpellier
Locations (1):
- University hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC